CLINICAL TRIAL: NCT04315506
Title: A Text-based Reduction Intervention for Smokeless Tobacco Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00103410
Record Dates: First submitted 2020-03-18; First posted 2020-03-19 (Actual); Results first posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Smokeless Tobacco Cessation
Keywords: smokeless tobacco; quitting smokeless tobacco
MeSH Terms: conditions — Tobacco Use Cessation; Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- #EnufSnuff.TXT Intervention (Experimental): Scheduled gradual reduction. Participants are asked to gradually reduce smokeless tobacco usage.
  Interventions: Behavioral: #EnufSnuff.TXT Intervention
- Enough Snuff Intervention (Active Comparator): Participants in this arm will be given the Enuff Snuff cessation manual.
  Interventions: Behavioral: Enough Snuff Intervention

INTERVENTIONS:
Behavioral: #EnufSnuff.TXT Intervention — The SGR program will reduce smokeless tobacco until you reach zero. The intent of this program is to reduce the number of times participants use smokeless tobacco down to zero. Participants will also receive text-based support messages.
  Arms: #EnufSnuff.TXT Intervention
Behavioral: Enough Snuff Intervention — Participants will be sent the Enough Snuff cessation manual. One weeks after it is sent, participants will then receive text messages from the study team twice a week for ten weeks.
  Arms: Enough Snuff Intervention

SUMMARY:
Participants will be randomly assigned (like the flip of a coin) to one of the two groups after completing the baseline survey. Participants have a 50% of being in either the #EnufSnuff.TXT intervention group or the Enough Snuff Intervention group. Participants will then be given a baseline survey and the intervention will be explained to them.

DETAILED DESCRIPTION:
Group 1: #EnufSnuff.TXT intervention For participants in the #EnufSnuff.TXT intervention, this program will occur for up to 10 weeks. The intent of this program is to reduce the number of times participants use smokeless tobacco to zero. Participants will also be provided with cessation support messages. During the first week, participants will be asked to use smokeless tobacco as per their regular habit. They will be required to text "s" every time they use smokeless tobacco . At the end of the week we will confirm how many times you dip a day on average. Based on this number participants will be texted a reduction schedule over the next several weeks to assist with cessation. During these weeks participants will be instructed not to use smokeless tobacco unless they receive a text message telling them to do so. Within 30 minutes after participants receive the text message, they will be required to respond to that message and text the study team "s" if they used smokeless tobacco. Participants will still be required to let the study team know if they used smokeless tobacco at a different time than the time we text participants. This will help the study team know if participants have followed the schedule or not. However, if the pattern continues then participants will receive a call from the study coordinator to reexamine their pattern of smokeless tobacco use and readjust your schedule.

Group 2: Enough Snuff Intervention group

Participants in the control group will be sent the Enough Snuff cessation manual. One week after it is sent, participants will then receive two text messages a week from the study for ten weeks. These messages will reference the cessation manual.

End of Intervention and 3 and 6 Month Follow-up Assessments For both study groups, participants will be asked to take a follow-up survey at end of program and 6 months after the baseline survey. At three months all participants will be sent a brief assessment about smokeless tobacco use via text. If participants have reported to the study team that they have quit using smokeless tobacco, a small percentage of participants may be asked to provide a saliva sample to check for nicotine.

ELIGIBILITY:
Inclusion Criteria:

* 1) 18 years of age and older
* 2) Have used smokeless tobacco for the last year, currently dip 3 or more times a day
* 3) Have an address in a rural census tract defined by a RUCC code of 4-10 and/or an IMU of 62 or lower
* 4) Interested in participating in a cessation program; and
* 5) Have access to a cell phone with unlimited texting ability.

Exclusion Criteria:

* 1) Non-English speaking;
* 2) Have smoked cigarettes or used any other tobacco product in the past 30 days (i.e., dual user) and are not willing to abstain during the intervention period
* 3) Currently participating in a smokeless tobacco cessation study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 532 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2023-01-28 (Actual); Study Completion 2023-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Devon Noonan, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Noonan D, Silva SG, Fish LJ, Simmons LA, Nwankwo N, Scherr K, Da Costa M, Sang E, Sanders C, Swinkels C, Garcia Ortiz N, Severson HH, Pollak KI. Randomized Controlled Trial of a Text-Based Smokeless Tobacco Cessation Intervention for Rural and Medically Underserved Communities. Nicotine Tob Res. 2024 Dec 23;27(1):132-142. doi: 10.1093/ntr/ntae182. PMID 39030750

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants recruited for the study using social media and other media advertisement outlets (i.e., Facebook, Instagram, Google Ads). An advertising profile for the study targeted the study population (e.g., smokeless tobacco users (chewer/dipper), over age 18, profiled for tobacco use) for rural and medically underserved counties in the U.S. This was a single- site study, which used electronic consents and survey measures.
Groups:
- #EnufSnuff.TXT Intervention: Scheduled gradual reduction. Participants are asked to gradually reduce smokeless tobacco usage.
  SGR: The SGR program will reduce smokeless tobacco use until you reach zero. The intent of this program is to reduce the number of times participants use smokeless tobacco down to zero. Participants will also receive text-based support messages.
- Enough Snuff Intervention: Participants in this arm will be given the Enuff Snuff cessation manual.
  Control: Participants will be sent the Enough Snuff cessation manual. One week after it is sent, participants will then receive text messages from the study team twice a week for ten weeks.
Period: Overall Study
Arm/Group | #EnufSnuff.TXT Intervention | Enough Snuff Intervention
Started | 264 | 268
Completed | 182 | 177
Not Completed | 82 | 91
Not completed — Lost to Follow-up | 74 | 82
Not completed — Withdrawal by Subject | 8 | 8
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | #EnufSnuff.TXT Intervention | Enough Snuff Intervention | Total
Number analyzed (Participants) | 264 | 268 | 532
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (11.9) | 45.1 (11.9) | 44.9 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 262 | 266 | 528
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 6 | 7
  Not Hispanic or Latino | 257 | 255 | 512
  Unknown or Not Reported | 6 | 7 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 257 | 255 | 512
  More than one race | 1 | 6 | 7
  Unknown or Not Reported | 6 | 7 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 264 | 268 | 532

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Did Not Use Chew/Dip in the Past 7 Days (Quit)
Description: Measured by self-report. Number of participants who replied "no" the following: "In the past 7 days, have you used chew/dip?- Yes or No".
Time Frame: 6 months post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | #EnufSnuff.TXT Intervention | Enough Snuff Intervention
Number analyzed (Participants) | 264 | 268
Participants | 61 | 56
Statistical Analysis 1: Comparison: #EnufSnuff.TXT Intervention vs Enough Snuff Intervention; Test type: Superiority; p = 0.5384, Regression, Logistic — The analysis was a two-intervention arm comparison. Adjustments for multiple tests and outcomes were not required; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.75 to 1.72] — Odds of quitting in Enuf Snuff group (SGR) compared to Enough Snuff (control)

2. Secondary Outcome: Change in Withdrawal as Measured by Minnesota Nicotine Withdrawal Scale (MNWS)
Description: The MNWS is a seven-item scale that measures withdrawal symptoms (i.e., irritability, anxiety, difficulty concentrating, restlessness, increased appetite or weight gain, depression, and insomnia) during the past 24 hours. Each item was measured using a Likert scale (with 0 = not present to 4 = severe). A nicotine withdrawal total score was derived by summing the scores for the 7-items, with a possible range from 0 to 28, and higher scores indicating greater withdrawal.
Time Frame: Baseline, 3 months, and 6 months post-randomization
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | #EnufSnuff.TXT Intervention | Enough Snuff Intervention
Number analyzed (Participants) | 264 | 268
score on a scale
  Baseline | 7.3 (6.3) | 7.1 (5.7)
  3 Months | 6.3 (5.2) | 5.9 (5.4)
  6 Months | 5.8 (5.8) | 5.4 (5.4)
Statistical Analysis 1: Comparison: #EnufSnuff.TXT Intervention vs Enough Snuff Intervention; For secondary outcomes, the study was not powered. The null hypothesis was no between-treatment arm difference in the trajectory of change from baseline to six months; Test type: Superiority; p = 0.6624, Mixed Models Analysis — P-value above is for the treatment-by-time squared term in the statistical model for longitudinal data; quadratic change in outcome determined, compared trajectory of outcome change in EnufSnuff (SGR) compared to Enough Snuff (control); Multi-level, mixed-effects model for longitudinal data was conducted; Slope = -0.1057, 95% CI 2-sided [-0.5808 to 0.3693] — Slope difference estimate reported above, estimate compares trajectory slope coefficient for EnufSnuff (SGR) to slope coefficient for Enough Snuff (control)

3. Secondary Outcome: Change in Craving as Measured by Smokeless Tobacco Evaluation Questionnaire (STEQ)
Description: The STEQ is a 12-item scale assessing the degree to which participants experience the reinforcing effects of smokeless tobacco on a 7-point Likert scale (0= not at all to 7=Extremely). The tool has five subscales: chewing satisfaction, psychological reward, enjoyment of sensations in cheek/gum, craving reduction, and aversion. To assess change in craving, the one item craving reduction subscale was used for this analysis. The question was "Did chewing/dipping immediately relieve your craving for smokeless tobacco?". The possible range was 0= not at all to 7=Extremely. At each timepoint, a higher score on this item indicated greater withdrawal symptom in terms of craving relief. Thus, a decrease in the mean craving reduction score across time indicates an improvement in the withdrawal symptoms specific to craving.
Time Frame: Baseline, 3 months, and 6 months post-randomization
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | #EnufSnuff.TXT Intervention | Enough Snuff Intervention
Number analyzed (Participants) | 264 | 268
score on a scale
  Baseline | 5.1 (1.6) | 5.1 (1.5)
  3 Months | 5.0 (1.5) | 4.8 (1.6)
  6 Months | 4.7 (1.6) | 4.6 (1.7)
Statistical Analysis 1: Comparison: #EnufSnuff.TXT Intervention vs Enough Snuff Intervention; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.2320, Mixed Models Analysis — A multi-level, mixed-effects model for longitudinal data was applied. The p-value provided above was for the treatment-by-time effect used to test for differences in the trajectory of change in craving reduction between the two treatment groups; Multi-level, mixed-effects model for longitudinal data was conducted. (trajectory analysis); Slope = .0946, 95% CI 2-sided [-0.0609 to 0.2501] — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | #EnufSnuff.TXT Intervention | Enough Snuff Intervention
All-Cause Mortality (participants affected / at risk) | 0/264 | 0/268
Serious Adverse Events (participants affected / at risk) | 0/264 | 0/268
Other Adverse Events (participants affected / at risk) | 0/264 | 0/268

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-01-28): https://cdn.clinicaltrials.gov/large-docs/06/NCT04315506/Prot_001.pdf
  • Statistical Analysis Plan (2022-01-28): https://cdn.clinicaltrials.gov/large-docs/06/NCT04315506/SAP_002.pdf
  • Informed Consent Form (2022-01-28): https://cdn.clinicaltrials.gov/large-docs/06/NCT04315506/ICF_000.pdf